CLINICAL TRIAL: NCT01306110
Title: Screening for Liver Fibrosis by Using Non-invasive Methods in Patients With Diabetes. A Prospective Study
Acronym: DIABSCAN
Status: Completed | Type: Observational
Sponsor: Association HGE CHU Bordeaux Sud (Other)
Responsible Party: Principal Investigator, de Ledinghen, Professor, Association HGE CHU Bordeaux Sud
Other Study IDs: FS02-062007
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes
Keywords: Liver fibrosis; diabetes; Fibroscan; Fibrotest; noninvasive fibrosis biomarkers
MeSH Terms: conditions — Diabetes Mellitus; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to evaluate liver fibrosis using FibroScan and biochemical markers in patients with diabetes.

DETAILED DESCRIPTION:
Patients with diabetes are at risk for nonalcoholic fatty liver disease (NAFLD) leading to advanced fibrosis, cirrhosis, and liver cancer. However, liver fibrosis screening in this large population needs non-invasive methods. Recently, FibroScan was shown to be a good method for the diagnosis of advanced fibrosis in NAFLD patients. We examined the efficacy of a screening strategy with a noninvasive fibrosis biomarker (FibroTest) and transient elastography (FibroScan) in patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects
* More than 18 years of age
* Patients with Diabetes
* Written informed consent

Exclusion Criteria:

* Patients refusing to participate to the study and to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetes
Sampling Method: Non-Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2007-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor De Ledinghen, MD PhD, Study Director — University Hospital, Bordeaux; Juliette Foucher, MD, Principal Investigator — University Hospital, Bordeaux; Julien Vergniol, MD, Principal Investigator — University Hospital, Bordeaux; Vincent Rigalleau, MD PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Service Hepato-Gastroentérologie Hopital Haut-Leveque, Pessac, France